CLINICAL TRIAL: NCT04960371
Title: Effects of Anxiety on Coronary Microcirculatory Function in Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018058
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Coronary Microvascular Disease; Anxiety State
Keywords: anxiety; coronary microcirculatory function; hypertension
MeSH Terms: conditions — Microvascular Angina; Anxiety Disorders; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anxiety group: the score of Self-rating Anxiety Scale greater than 50
  Interventions: Diagnostic Test: coronary flow reserve (CFR)
- non-anxiety group: the score of Self-rating Anxiety Scale less than 50
  Interventions: Diagnostic Test: coronary flow reserve (CFR)

INTERVENTIONS:
Diagnostic Test: coronary flow reserve (CFR) — Coronary flow velocity profiles in the left anterior descending artery were obtained using colour-guided pulse wave Doppler. We measured peak diastolic coronary flow velocity of the diastolic coronary waveform at rest and after ATP infusion (140 µg/kg. min) for 2 min. The CFR was calculated as the ratio of hyperaemic peak diastolic velocity to resting baseline diastolic velocity. All patients abstained from caffeine-containing drinks for at least 24h before testing.

SUMMARY:
This study assessed anxiety status and coronary flow reserve in hypertensive patients to investigate the effects of anxiety on coronary microcirculatory function.

DETAILED DESCRIPTION:
This study assessed anxiety status and coronary flow reserve in hypertensive patients to investigate the effects of anxiety on coronary microcirculatory function.The hypertensive patients with chest pain for suspicious coronary heart disease were seriesly enrolled. All the patients underwent coronary angiography or coronary CT angiography to exclude the diagnosis of obstructive coronary artery disease . Coronary flow reserve (CFR) is an integrated measure of flow through both the large epicardial arteries and the coronary microcirculation. In the absence of obstructive stenosis of the epicardial arteries, CFR is an indicator of coronary microcirculatory function，which can be assayed by Transthoracic Doppler echocardiography. The symptoms of anxiety were measured with Self-rating Anxiety Scale (SAS) . According to the SAS score,the patients were divided into anxiety group and non-anxiety group.We assessed the association of anxiety with coronary microcirculatory function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clear diagnosis of hypertension (≥1 year, drug control within 140/90mmHg); (2) Significant coronary artery stenosis was excluded by imaging within 1 year (≤50%); (3) Age between 18 and 80.

Exclusion Criteria:

1. CHD, heart valve disease, congenital heart disease, cardiomyopathy and pericardial disease; (2) Left ventricular ejection fraction (LVEF) <50%; (3) Increased markers of myocardial injury; (4) Diabetes mellitus, connective tissue disease, chronic obstructive pulmonary disease and malignant tumor; 5) Severe hepatic and renal impairment (Cr ≥120 umol/L, ALT ≥120 umol/L); 6) Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The hypertensive patients with chest pain for suspicious coronary heart disease (CHD) in Peking University Third Hospital were seriesly enrolled. All the patients underwent coronary angiography or coronary CT angiography to exclude the diagnosis of OCAD.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Coronary flow reserve | baseline
  Coronary flow reserve (CFR) is an integrated measure of flow through both the large epicardial arteries and the coronary microcirculation. In the absence of obstructive stenosis of the epicardial arteries, CFR is an index of coronary microcirculatory function.

SECONDARY OUTCOMES:
Inflammatory mediators | baseline
  Inflammatory mediators were measured using Quantibody Human Immune Response Array.

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Guo, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No